CLINICAL TRIAL: NCT03682367
Title: Perioperative Analgesia Using Gabapentin in Head and Neck Cancer Surgery: A Randomized Controlled Trial
Brief Title: Perioperative Analgesia Using Gabapentin in Head and Neck Cancer Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor Recruitment
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1166778
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Cancer of Head and Neck; Narcotic Use
Keywords: Gabapentin; Narcotic; Cancer; Placebo
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All staff involved including nursing, surgeons, pain management, participants and PI will be blinded. Unmasked personnel only include research pharmacy staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Standard of care use of perioperative analgesia with acetaminophen and opioids that is supplemented with placebo solution. Participants will then be discharged after surgery with postoperative acetaminophen, opioids, and placebo.
  Interventions: Drug: Placebo - Concentrate
- Intervention (Experimental): Interventional use of perioperative analgesia with acetaminophen and opioids that is supplemented with gabapentin solution. Participants will then be discharged after surgery with postoperative acetaminophen, opioids, and gabapentin.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Use of Gabapentin peri- and post-operatively.
  Other Names: Neurontin; Gralise; Horizant
  Arms: Intervention
Drug: Placebo - Concentrate — Use of sugar-free Placebo peri- and post-operatively.
  Arms: Control

SUMMARY:
Patients undergoing head and neck cancer surgery often have a lot of pain after surgery, which can lead to a need for a lot of narcotic pain medication. These medications can have many side effects that can make recovery more difficult including nausea, vomiting, dizziness, being overly sleepy, itchiness, inability to urinate, confusion, inability to have a bowel movement, longer time before being able to start walking. These side effects can make the hospital stay longer. The use of gabapentin, which is a non narcotic pain medication that focuses on nerve pain, has been used in smaller head and neck surgeries including removal of tonsils, sinus surgery, thyroid surgery. Studies in patients needing orthopedic or OB/Gyn surgery have shown improved pain control with gabapentin. Potential benefits to future patients include improved pain control, less narcotic associated side effects and faster functional recovery.

DETAILED DESCRIPTION:
Patients undergoing head and neck cancer surgery frequently experience significant post surgical pain, which often necessitates the use of narcotic pain medication. However, opioids can have multiple side effects that can complicate the head and neck cancer surgery patients postoperative care including nausea, vomiting, dizziness, sedation, pruritis, urinary retention, delirium, constipation, and time to ambulation. This, in turn, may affect patient length and cost of hospital stay. Consequently, a multimodal approach to analgesia is often employed with a focus on use of scheduled acetaminophen +/- NSAIDs supplemented with narcotics.

The use of gabapentin in the head and neck surgery literature has largely been limited to outpatient surgeries, including tonsillectomy in children and adults, functional endoscopic sinus surgery, and thyroidectomy. Indeed, a recent systematic review examined RCT comparing multimodal analgesia with gabapentin to analgesia without gabapentin in the otolaryngology literature. The majority of these studies employed preoperative dosing only, with only 1 study providing a single postoperative dose as well. The control group pain regimen among these studies did vary and included a combination of acetaminophen, NSAIDs, dexmedetomidine, or clonidine supplemented with opioids. The studies focused on the impact of gabapentin on acute postoperative pain determined by subjective measurement of reduction in visual analog pain scale. Of note, these patients were not hospitalized for longer than 24 hours. The thyroid and sinus studies consistently demonstrated improved pain control with use of gabapentin compared to control. The data was slightly more variable across the tonsillectomy studies. Moreover, 7 studies also measured the need for breakthrough pain medication and supplemental analgesia; each of these studies demonstrated significantly less supplemental analgesia consumption in the gabapentin group.

The only study examining the utility of gabapentin in pain management in head and neck cancer patients (glossectomy with anterolateral thigh free flap) examined the utility of a single preoperative dose. The authors concluded that this led to a significant reduction in subjective postoperative pain scores, morphine requirement, and nausea and vomiting compared to controls. This study did not employ postoperative gabapentin.

Furthermore, a recent meta analysis (133 RCT) examining literature across multiple surgical specialties pertaining to the efficacy of perioperative gabapentin supplementation vs placebo. The meta analysis indicated both the efficacy of gabapentin supplementation in decreasing opioid requirement (measured via morphine equivalent units) in the experimental group during the first 24 hours (P<0.001), as well as a good safety profile across a wide range of loading and maintenance doses (200 to 1200 mg) of gabapentin. The significant reduction in opioid requirement was independent of surgery type. Moreover, the gabapentin group demonstrated a significant decrease in VAS postoperative pain scores, nausea, vomiting and itching; however, sedation scores were increased. Only 8 of these 133 RCT examined the effect of gabapentin outside the immediate 24 hour period, and all 8 trials demonstrated improvement in chronic pain scores at 3 months post-operatively. Finally, patient satisfaction scores and preoperative anxiety were also significantly improved with the use of gabapentin compared to controls.

Here, the investigators propose, for the first time, a superiority double blind randomized controlled placebo trial examining the effect of perioperative supplementation with gabapentin in head and neck cancer patients undergoing surgery. The primary purpose of this study is to determine the difference in morphine equivalent units between the experimental (i.e. perioperative gabapentin) and control group (i.e. no perioperative gabapentin). The secondary purpose of this study is to determine differences across the two groups in relation to the following: visual analog pain scores, cost and length of stay, medication side effects, and incidence of postoperative complications. Of note, in order to maximize reliability of the visual analog scale (VAS), prior studies have employed the Jadad scoring system, which the investigators will also implement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major head and neck surgery with concomitant free flap reconstruction surgery at UCDMC (oncology and non-oncologic): There will be two groups. Group 1 will include reconstruction with fibula free flap only. Group 2 will include any other free flap reconstruction, including scapular free flap, radial forearm free flap, anterolateral thigh free flap, anteromedial thigh free flap, and latissimus dorsi free flap.
* Patients naïve to gabapentin
* Adult patients >18 years of age and able to consent

Exclusion Criteria:

* Patients who are already taking scheduled gabapentin
* Patients allergic to gabapentin
* Chronic opioid use not from active head and neck cancer
* Illicit drug use (per report)
* Patients with known renal compromise, such that Creatinine clearance is < 30
* Patient with known hepatic insufficiency or cirrhosis
* Adults unable to consent
* Individuals less than 18 years old
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bewley, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 4 | 4
Completed | 2 (Withdrawn due to non-compliance) | 0 (Patients withdrawn due to confounding neuropathic pain or exited early from study.)
Not Completed | 2 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Closed Study Early | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Morphine Equivalent Units
Description: Determine the difference in average morphine equivalent units between experimental and control group.
Time Frame: Perioperative.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Average Morphine Equivalent Units
Description: Determine the difference in average morphine equivalent units between experimental and control group.
Time Frame: 1 week post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Average Morphine Equivalent Units
Description: Determine the difference in average morphine equivalent units between experimental and control group.
Time Frame: 30 days post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Score (10 Point VAS)
Description: Determine average change of inpatient Pain Score Visual Analog Scale (VAS) on a standardized 1 (no pain) to 10 (highest level of pain) scale between experimental and control groups.
Time Frame: Perioperative, 1 week post-operation, 1 week post-discharge, and 30 days post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Post-operative Complications
Description: Incidence of postoperative complications between experimental and control group.
Time Frame: 30 days post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Narcotics-related Complications
Description: Incidence of narcotics-related complications between experimental and control group.
Time Frame: 30 days post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Inpatient Length of Stay
Description: Determine the difference of average inpatient length of stay between experimental and control group.
Time Frame: 1 week post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Inpatient Cost
Description: Determine the difference of average inpatient cost between experimental and control group.
Time Frame: 1 week post-operation.
Population: Due to safety concerns and patient non-compliance, the data was unreliable and uninterpretable.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Any known untoward event of any severity that occurs subsequent to the AE reporting period that the Investigator assesses as at least possibly related to the study therapy (i.e., the relationship cannot be ruled out) should also be reported as an AE.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=4) | Intervention (N=4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Constipation
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea

LIMITATIONS AND CAVEATS:
Early study termination was decided after several technical issues regarding study logistics and patient non-compliance lead to unreliable and uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03682367/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03682367/ICF_001.pdf